CLINICAL TRIAL: NCT06511037
Title: The Impact of Pafolacianine Injection for Intraoperative Imaging on Outcomes of Gastrointestinal Cancer Peritoneal Carcinomatosis - A Pilot Study
Brief Title: PhI Pilot Study Pafolacianine Inject for Intraoperative Imaging on Outcomes of GI Cancer Peritoneal Carcinomatosis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: On Target Laboratories (Unknown)
Responsible Party: Principal Investigator, Maheswari Senthil, MD, Professor of Surgery, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4951; UCI 23-184 (Other: UCI CFCCC)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Gastrointestinal Cancer; Peritoneal Carcinomatosis
MeSH Terms: conditions — Gastrointestinal Neoplasms; Peritoneal Neoplasms | interventions — Pafolacianine; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pafolacianine (CYTALUX) (Experimental): All subjects will receive one single intravenous infusion of 0.025 mg/kg of pafolacianine (CYTALUX) injection prior to anticipated intraoperative imaging planned for cytoreductive surgery.
  Interventions: Drug: Pafolacianine (CYTALUX) with intraoperative fluorescent near-infrared (NIR) imaging

INTERVENTIONS:
Drug: Pafolacianine (CYTALUX) with intraoperative fluorescent near-infrared (NIR) imaging — Given IV

SUMMARY:
This is a pilot, single-arm, open label study to evaluate the ability of CYTALUX™ (pafolacianine) to help identify cancerous lesions in subjects with gastrointestinal cancers and peritoneal carcinomatosis during cytoreductive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age and older
* Have a primary diagnosis of primary gastrointestinal cancer (of adenocarcinoma), planned for cytoreductive surgery
* Female patients must have a negative serum pregnancy test at screening, followed by a negative urine pregnancy test on the day of scheduled study drug infusion, or day of surgery
* Female patients of childbearing potential, or less than two (2) years postmenopausal, agree to use an acceptable form of contraception from time of signing informed consent until 30 days after study completion
* Ability to understand the requirements of the study, provide written informed consent for participation in the study and authorization of use and disclosure of protected health information, and agree to abide by study restrictions

Exclusion Criteria:

* Previous exposure to CYTALUX™ (PAFOLACIANINE)
* Patients with known gastrointestinal cancer with carcinomatosis determined pre-operatively to be inoperable
* Any medical condition that in the opinion of the investigators could potential jeopardize the safety of the patient
* History of anaphylactic reaction
* History of allergy to any components of CYTALUX™ (PAFOLACIANINE), including folic acid
* Pregnancy, or positive pregnancy test
* Clinically significant abnormalities on ECG
* Impaired renal function defined as eGFR <50 mL/min/1.73m2
* Impaired liver function defined as values >3x the upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin
* Received an investigational agent in another trial within 30 days prior to surgery
* Known sensitivity to fluorescent light

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Cytoreduction (CC) Score | 1 year
  Describe the completeness of cytroreduction (cc) score with Cytoreductive surgery (CRS) with Cytalux injection.
Sensitivity-True Positive Rate (TPR) | 1 year
  Sensitivity, or the True Positive Rate (TPR), is defined as the proportion of fluorescent light positive lesions that are histologically confirmed to be gastrointestinal cancer (and folate receptor (FR) positive) by central pathology relative to the total number of lesions confirmed to be gastrointestinal cancer (FR+) by central pathology, that is proportion of cancerous lesions that are fluorescent light positive.
Specificity-True Negative Rate (TNR) | 1 year
  Specificity, or the True Negative Rate (TNR), is defined as the proportion of fluorescent light negative lesions that are histologically negative for gastrointestinal cancer and FR- by central pathology, relative to the total number of lesions that are negative for gastrointestinal cancer (FR-) by central pathology-that is, the proportion of non-cancer lesions that are fluorescent light negative.
Positive Predictive Value (PPV) | 1 year
  Positive Predictive Value (PPV) is defined as the proportion of fluorescent light positive lesions that are histologically confirmed to be FR+ and gastrointestinal cancer by central pathology relative to the total number of lesions removed that are fluorescent light positive-that is, the proportion of fluorescent light positive lesions that are cancerous.
Negative Predictive Value (NPV) | 1 year
  Negative Predictive Value (NPV) is defined as the proportion of fluorescent light negative lesions that are histologically negative for gastrointestinal cancer and FR- by central pathology relative to the total number of lesions removed that are fluorescent light negative-that is, the proportion of fluorescent light negative lesions that are histologically negative for cancer.
Accuracy | 1 year
  Accuracy is defined as the proportion of fluorescent light positive lesions that are histologically confirmed to be FR+ and gastrointestinal cancer by central pathology and the fluorescent light negative lesions that are histologically negative for gastrointestinal cancer and FR- by central pathology relative to all lesions sampled.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 30 days
  Incidence rates of all treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) from the time of CYTALUX (PAFOLACIANINE) injection administration through the conclusion of study participation

CONTACTS AND LOCATIONS:
Overall Officials: Maheswari Senthil, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No